CLINICAL TRIAL: NCT03700255
Title: Efficacy of a Simulator Based (PickUpSimTM) Residents' Training Program for Oocyte Retrievals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/03
Record Dates: First submitted 2018-09-24; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Infertility; Oocytes; Fertilization in Vitro
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will undergo the PickUpSimTM simulation training program
  Interventions: Procedure: PickUpSimTM simulation training program
- Group B (No Intervention): Group B will only have the classic training with no simulation.

INTERVENTIONS:
Procedure: PickUpSimTM simulation training program — The residents will take part in simulation sessions of 30 minutes duration. There will be 4 training sessions with seven simulation scenarios available. During the sessions, the following data will be collected for each scenario success or failure, reason for failure, time needed for completion, and oocyte retrieval rate. All scenarios will be repeated in the same conditions in the second week and data collected again. In the following 15 days, residents will start performing OPU, under direct supervision from senior physicians. For each patient, the resident will puncture one ovary. During the retrieval, the operator will specify the number of follicles punctured for each collected tube. The identity of the operator and the number of follicles punctured (per tube and in total) are noted on a separate sheet entitled the "retrieval sheet". After the first month, residents will start performing all the OPUs, including both ovaries, supervised by the senior physicians.
  Arms: Group A

SUMMARY:
Simulation is an educational approach that has recently found an application in healthcare.acquire. Angers university hospital has decided to acquire, in December 2016, the high-fidelity Oocyte Pick up (OPU) simulator PickUpSimTM, and the investigators have put in place a training novel program containing different simulation based courses. It is essential to analyze its impact on the clinical practice before implementing it on a larger scale. Initial hypothesis was that the residents' lack of specific training and inexperience would result in suboptimal oocyte retrievals, especially for their first cases

The investigators will undertake a prospective comparative study at the In Vitro Fertilization (IVF) unit of the Angers University Hospital between May 2019 and April 2022. The investigators will include all voluntary residents in rotation at the IVF unit in that time period. The participants will be divided in two groups: Group A will undergo the PickUpSimTM simulation training program whereas group B will only have the classic training with no simulation.

The primary objective is to assess the benefits of an OPU simulation training program using the PickUpSimTM simulator for teaching residents in a university-affiliated IVF center. The main criterion the investigators will use is the "oocyte retrieval rate" (ORR) during the first month following 15 days of simulation training. The ORR is calculated as the number of oocytes retrieved divided by the number of follicles aspirated.

Our secondary objectives are:

* To assess the residents' satisfaction with the simulation training program.
* To evaluate the learning curve of residents during the two weeks of training.
* To compare the OPU complication rate between residents with and without previous simulation training.
* To analyze the oocyte retrieval rate in the second and third month of REI rotation for residents, and compare it between those with and those without simulation training.

DETAILED DESCRIPTION:
Hypotheses and Objectives The initial hypothesis was that the residents' lack of specific training and inexperience would result in suboptimal oocyte retrievals, especially for their first cases. This could potentially decrease the overall success rates of a university-affiliated IVF unit (a lower oocyte yield would lead to a lower number of embryos, thus decreasing pregnancy and live birth rates). The investigators aim to analyze whether residents who had previous OPU simulation training would have better oocyte retrieval rates than residents without pervious simulation training.

1. Primary objective The primary objective is to assess the benefits of an OPU simulation training program using the PickUpSimTM simulator for teaching residents in a university-affiliated IVF center. The main criterion is the "oocyte retrieval rate" (ORR) during the first month following 15 days of simulation training. The ORR is calculated as the number of oocytes retrieved divided by the number of follicles aspirated.
2. Secondary objectives

The secondary objectives are:

* To assess the residents' satisfaction with the simulation training program.
* To evaluate the learning curve of residents during the two weeks of training.
* To compare the OPU complication rate between residents with and without previous simulation training.
* To analyze the oocyte retrieval rate in the second and third month of REI rotation for residents, and compare it between those with and those without simulation training.

The investigators will use the following tools to analyze the secondary objectives:

* A survey filled by residents at the end of the first month of REI rotation. The first part of the survey covers all aspects of the simulation training sessions (number and duration, quality of scenarios, similarity to real life events), and will be completed only by the residents who had the training sessions. However, the second part of the survey includes questions about the residents' impressions while performing their first oocyte retrievals on actual patients (stress levels, self-confidence…), and will be completed by all residents.
* Analysis of data collected from the training sessions with PickUpSimTM. There are seven scenarios in the training program, and each resident will complete each scenario twice. For each scenario, the data collected will include: success or failure, reason for failure, time needed for completion, and oocyte retrieval rate. Information will be analyzed per resident in order to assess whether the competence level improves with training.
* Collection and analysis of information regarding postoperative complications. Postoperative complications are defined as a hemoperitoneum requiring a surgical intervention, or infections requiring antibiotic therapy or a surgical intervention, occuring in the month following the OPU.
* The oocyte retrieval rate of residents who had simulation training and those who did not in the second and third month of REI rotation.

Methodology / Study diagram

The investigators will undertake a prospective comparative study at the IVF unit of the Angers University Hospital between May 2019 and April 2022. The investigators will include all residents in rotation at the IVF unit in that time period. The residents can decide whether or not to partake in the study. Participants will be divided in two groups: Group A will undergo the PickUpSimTM simulation training program whereas group B will only have the classic training with no simulation. The group allocation will be based on the timing of the REI rotation: Residents rotating between May and November will be assigned to group A and those rotating between November and May will be assigned to group B. In France, obstetrics and gynecology residents switch rotations every semester (6 months), for a total period of training of 5 years (10 semesters). Residents choose their own rotations, with minimum requirements to obtain the national diploma. For instance, one semester in an REI department is required for the obstetrics and gynecology diploma. Moreover, residents in "medical gynecology" and "endocrinology" also have a 6 months rotation in an REI department. Most often, residents choose the REI rotation towards the end of their training, in their last two years. We will include in our study all residents rotating in the REI department (2 to 3 per semester), regardless of their diploma or the year of training.

1. Simulation training program of group A

   During the first 15 days of their REI rotation, residents will observe all OPU performed by the department's senior physicians in the operating room, usually early in the morning. Later during the day, the residents will take part in simulation sessions of 30 minutes duration, led by the same physician who performed the retrievals in the morning. There will be a total of 4 training sessions, two sessions the first week, and two sessions the second. The seven simulation scenarios available will be played out during the first week, three in the first training session and four in the second. The chronological order of scenarios will be randomly decided by the supervising physicians. During the sessions, the following data will be collected for each scenario : success or failure, reason for failure, time needed for completion, and oocyte retrieval rate. All scenarios will be repeated in the same conditions during the two sessions in the second week and data collected again. Six different senior gynecologists will supervise the simulation sessions: 3 attending physicians (Dr. Bouet, Dr. Dreux and Dr. Jeanneteau), and 3 senior REI fellows (Dr. Faurant, Dr. Abnoun, and Dr. Delbos).

   In the following 15 days, residents will start performing OPU, under direct supervision from senior physicians. For each patient, the resident will puncture one ovary and the senior the other. The choice of sides will not be predefined, but will be decided by the attending and resident immediately before the procedure. A transvaginal ultrasound will be performed to assess the feasibility of the retrieval and the accessibility of the ovaries. If both ovaries are easily accessible, the decision will be made by mutual consent. If one side is deemed more difficult, it will be handed to the senior.

   During the retrieval, the operator will specify the number of follicles punctured for each collected tube. The operating room nurse will assign a number to each tube (1, 2, 3…) and register on a separate paper the number of tubes and number of follicles aspirated per tube. When one side is completed, and before changing operators, the aspiration tubing is flushed and the content is added to the last tube, since some oocytes may be stuck in the tubing. The same procedures are repeated for the second operator (tube numbers, number of follicles, flushing). The identity of the operator and the number of follicles punctured (per tube and in total) are noted on a separate sheet entitled the "retrieval sheet" (annex 3). Difficulties or incidents encountered during the retrieval are also noted. The tubes are then passed in a specific container at 37°C to the IVF laboratory, where the biology technicians will check the follicular fluid for oocytes. The retrieval sheet is handed along with the container.

   At the end of the first month of REI rotation, the residents will fill a 15 question survey to evaluate their satisfaction with the simulation training program, and their impressions while performing their first retrievals on patients . After the first month, residents will start performing all the OPUs, including both ovaries, supervised by the senior physicians, who will only intervene in difficult cases. Any senior intervention will be noted on the retrieval sheets. The same procedures and data collection will be conducted until the end of the semester.
2. Training program of Group B During the first 15 days of rotation, the residents will only observe the seniors performing the retrievals in the operating room. Since there is no simulation training, they will start performing OPU immediately after the observation period. The OPU procedures and the data collection will be the same as in Group A (One ovary first, tube numbers, number of follicles…). At the end of the first month, the residents will fill the survey regarding their impressions during their first retrievals . Following the first month, the residents start performing the entire retrievals, supervised by seniors who only intervene in difficult cases. Residents in group B can still use PickUpSimTM if they want to, but only after the first month and supervised by physicians.

Inclusion and exclusion criteria

1. Inclusion criteria All residents starting their REI rotation at the IVF center at Angers University Hospital between May 2018 and November 2020 will be included.
2. Exclusion criteria

   * Residents who refuse to partake in the study.
   * Residents who have already performed OPU during their residency training.
   * Retrieval sheets missing any kind of information (number of tubes or follicles, absent identification…).
   * Difficult OPU cases that end up being performed entirely by the senior physician (difficult visualization or access, mobile ovaries…).

Cases where the retrieval on one side is started by the resident but completed by the senior physician will not be excluded, since we aim to perform an intention-to-treat analysis. We will secondarily perform a per-protocol analysis, where these retrievals will be excluded.

Material The simulation training will be performed on PickUpSimTM. It is a high-fidelity simulator for oocyte retrievals, developed by the company ACCURATE, and costing 20 000€.

PickUpSimTM has several benefits. First of all, it has a haptic feedback system that allows the user to experience the resistance to penetration of the soft tissues, such as the ovarian surface and the follicle wall resistance. It also has a virtual transvaginal echographic monitor, and an ultrasound probe that can be rotated and moved in the transverse and sagittal planes, allowing the user to explore the ovary and the surrounding tissues (blood vessels, bowel loops…) in order to choose the best and safest entry plane for the retrieval. The simulator allows for forward and backward movement of the needle, and permits simulation of follicle emptying (with the use of a pedal pump) as well as flushing. The simulation scenarios are based on real clinical images, and allow for a precise evaluation of the trainee's performance, taking into account the proper movements to reach the desired follicles, the proper suction and washing technique and time, and the avoidance of the critical anatomical structures surrounding the ovary, such as blood vessels.

The simulation system is connected to a computer with an intuitive control software that allows the user to modify the settings. For instance, the user can change the aspiration pressure, add or remove the option of flushing the follicle, choose to activate aspiration via the foot pedal or the computer, change the caliber of the needle, and even modify the physics of the environment and the visibility of the needle in order to create more challenging scenarios.

ELIGIBILITY:
Inclusion Criteria:

* All voluntary residents starting their REI rotation at the IVF center at Angers University Hospital between May 2018 and November 2020 will be included.

Exclusion Criteria:

* Residents who refuse to partake in the study.
* Residents who have already performed OPU during their residency training.
* Retrieval sheets missing any kind of information (number of tubes or follicles, absent identification…).
* Difficult OPU cases that end up being performed entirely by the senior physician (difficult visualization or access, mobile ovaries…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
oocyte retrieval rate during the first month following 15 days of simulation training. | 6 month
  The ORR is calculated as the number of oocytes retrieved divided by the number of follicles aspirated

SECONDARY OUTCOMES:
the residents' satisfaction with the simulation training program | 6 month
  A survey filled by residents at the end of the first month of REI rotation
evaluate the learning curve of residents during the two weeks of training. | 6 month
  Analysis of data collected from the training sessions with PickUpSimTM. There are seven scenarios in the training program
compare the OPU complication rate between residents with and without previous simulation training | 6 month
  Collection and analysis of information regarding postoperative complications. Postoperative complications are defined as a hemoperitoneum requiring a surgical intervention, or infections requiring antibiotic therapy or a surgical intervention, occuring in the month following the OPU
the oocyte retrieval rate in the second and third month of REI rotation for residents | 6 month
  • The oocyte retrieval rate of residents who had simulation training and those who did not in the second and third month of REI rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers university hospital, Angers, France